CLINICAL TRIAL: NCT01284062
Title: A Phase 2a, Randomized, Double-blind, Sponsor Unblinded, Placebo-controlled, Multiple Dose Study To Evaluate The Pharmacodynamics, Pharmacokinetics And Safety Of Anrukinzumab In Subjects With Active Ulcerative Colitis
Brief Title: Pharmacokinetics/Pharmacodynamics Biomarker Study in Active Ulcerative Colitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B2421003; IMA-638 Anti-IL13 mAb; 2010-023762-49 (EudraCT Number)
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Colitis, Ulcerative
Keywords: Active Ulcerative Colitis; Phase 2A; Double-blind; Randomized; PK/PD Biomarker Study
MeSH Terms: conditions — Colitis, Ulcerative | interventions — anrukinzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): 200 mg PF-05230917, Anrukinzumab active dose level
  Interventions: Biological: Anrukinzumab
- Arm 2 (Experimental): 400 mg PF-05230917, Anrukinzumab active dose level
  Interventions: Biological: Anrukinzumab
- Arm 3 (Experimental): 600 mg PF-05230917, Anrukinzumab active dose level
  Interventions: Biological: Anrukinzumab
- Arm 4 (Placebo Comparator): Matching placebo - administered at matching dose level 200 mg, 400 mg or 600 mg.
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Anrukinzumab — 200 mg sterile liquid vial, administered intravenously, one-hour infusion on Day 1, Week 2, 4, 8, and 12
  Other Names: PF-05230917
  Arms: Arm 1
Biological: Anrukinzumab — 200 mg sterile liquid vial, dose level 400 mg administered intravenously, one-hour infusion on Day 1, Week 2, 4, 8, and 12
  Other Names: PF-05230917
  Arms: Arm 2
Biological: Anrukinzumab — 200 mg sterile liquid vial, dose level 600 mg administered intravenously, one-hour infusion on Day 1, Week 2, 4, 8, and 12 Note: dosing in the 600 mg arm will be delayed until the safety of the 200 mg and 400 mg arms has been reviewed.
  Other Names: PF-05230917
  Arms: Arm 3
Other: placebo — 200 mg liquid sterile vial, administered at matching dose level 200 mg, 400 mg or 600 mg intravenously, one-hour infusion on Day 1, Week 2, 4, 8, and 12
  Arms: Arm 4

SUMMARY:
This study represents the first investigation of anrukinzumab in patients with active ulcerative colitis (UC) and will evaluate proof of mechanism by changes in the mechanism based biomarker (YKL 40) and pharmacodynamic biomarkers (fecal calprotectin, lactoferrin and hs-CRP). It will provide further assessment of the safety, tolerability, and pharmacokinetics (PK) by administration of multiple intravenous (IV) doses of anrukinzumab.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, Age >=18 and <=65 years
* Active ulcerative colitis (UC) beyond the rectum based upon Mayo Score
* women of childbearing potential with highly effective method of contraception

Exclusion Criteria:

* Indeterminate disease status, Crohn's disease, ischemic colitis, positive HIV, positive or history of tuberculosis infection, active enteric infections, transplant organ recipient, concomitant steroids, immunosuppressives or anti-TNFs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (76):
- United States (48):
  - The Kirkland Clinic, Birmingham, Alabama
  - UAB Hospital, Birmingham, Alabama
  - UAB Hospital Department of Pharmacy, Birmingham, Alabama
  - Administrative Offices, Birmingham, Alabama
  - UAB ACIP, Birmingham, Alabama
  - Arizona Surgical Center, Phoenix, Arizona
  - Dedicated Phase I, Inc., Phoenix, Arizona
  - AGMG Endoscopy Center, Anaheim, California
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - West Coast Radiology Center, Santa Ana, California
  - Endoscopy Center of Connecticut, LLC, Hamden, Connecticut
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - International Clinical Research - US, LLC, Sanford, Florida
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - GI Diagnostics, Marietta, Georgia
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - Gastrointestional Associates, PA, Jackson, Mississippi
  - St. Dominic Hospital, Jackson, Mississippi
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - North Mississippi Medical Center, Tupelo, Mississippi
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Piedmont Gastroenterology Specialists, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center - Division of Gastroenterology and Liver Disease, Cleveland, Ohio
  - Wheeler and Stuckey, Inc., Oklahoma City, Oklahoma
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - OU Physicians Building, Oklahoma City, Oklahoma
  - Memphis Gastroenterology Group, PC, Germantown, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Centennial Medical Center Physicians Park, Nashville, Tennessee
  - Centennial Medical Center Tower Medical Imaging, Nashville, Tennessee
  - Columbia Medical Group - The First Clinic Inc., Nashville, Tennessee
  - Radiology Alliance, Nashville, Tennessee
  - Professional Quality Research, Inc., Austin, Texas
  - Austin Endoscopy Center, Austin, Texas
  - Austin Gastroenterology, PA, Austin, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Austin Gastroenterology, PA, Round Rocks, Texas
  - Cardiology Clinic of San Antonio, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - San Antonio Endoscopy Center, San Antonio, Texas
  - CNS Pharmacy, Murray, Utah
  - RGL Medical Services, Salt Lake City, Utah
  - Alpine Medical Group, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Wasatch Endoscopy Center, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
- Austria (3):
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Landesklinikum St. Poelten, Sankt Pölten
  - AKH Wien Universitaetsklinik fuer Innere Medizin III, Vienna
- Bulgaria (3):
  - MBAL Ruse / MHAT Ruse, Terapevtichno, gastroenterologichno i hematologichno otdelenie, Rousse
  - MBAL Voennomeditsinska Akademia / MMA HAT, Klinika po gastroenterologia i hepatologia, Sofia
  - DKTs Sveta Anna, Gastroenterologichen cabinet, Sofia
- Canada (5):
  - Heritage Medical Research Clinic - University of Calgary, Calgary, Alberta
  - Vancouver Coastal Health - Vancouver General Hospital, Vancouver, British Columbia
  - Vancouver General Hospital - The Gordon and Leslie Diamond Centre, Vancouver, British Columbia
  - The Religious Hospitallers of St. Joseph of the Hotel Dieu of Kingston, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- France (3):
  - CHU Hopital Nord, Amiens
  - Hopital Beaujon, Clichy
  - CHU Hotel-Dieu, Nantes
- Germany (4):
  - Charite - Campus Berlin Mitte, Berlin
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
- Hungary (3):
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak/I. Belgyogyaszati-Gasztroenterologiai Osztaly, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Clinfan Kft., Szekszárd
- Netherlands (3):
  - VU Medisch Centrum, Amsterdam
  - Academic Medical Center - University of Amsterdam, Dept. of Gastroenterology, Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
- Centralny Szpital Kliniczny MSWiA, Klinika Chorob Wewnetrznych i Gastroenterologii, Warsaw, Poland
- Sectia Clinica Medicina Interna II, Bucharest, Romania
- Spain (2):
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid

REFERENCES:
- [Derived] Reinisch W, Panes J, Khurana S, Toth G, Hua F, Comer GM, Hinz M, Page K, O'Toole M, Moorehead TM, Zhu H, Sun Y, Cataldi F. Anrukinzumab, an anti-interleukin 13 monoclonal antibody, in active UC: efficacy and safety from a phase IIa randomised multicentre study. Gut. 2015 Jun;64(6):894-900. doi: 10.1136/gutjnl-2014-308337. Epub 2015 Jan 7. PMID 25567115
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2421003&StudyName=Pharmacokinetics/Pharmacodynamics%20Biomarker%20Study%20in%20Active%20Ulcerative%20Colitis%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to anrukinzumab (PF-05230917) intravenous infusion over 1 hour on Day 1, Week 2, 4, 8 and 12.
- Anrukinzumab 200 mg: Anrukinzumab (PF-05230917) 200 milligram (mg) intravenous infusion over 1 hour on Day 1, Week 2, 4, 8 and 12.
- Anrukinzumab 400 mg: Anrukinzumab (PF-05230917) 400 mg intravenous infusion over 1 hour on Day 1, Week 2, 4, 8 and 12.
- Anrukinzumab 600 mg: Anrukinzumab (PF-05230917) 600 mg intravenous infusion over 1 hour on Day 1, Week 2, 4, 8 and 12.
Period: Overall Study
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Started | 21 | 21 | 21 | 21
Completed | 10 | 13 | 15 | 7
Not Completed | 11 | 8 | 6 | 14
Not completed — Adverse Event | 4 | 5 | 0 | 5
Not completed — Lack of Efficacy | 3 | 2 | 2 | 1
Not completed — Medication error without adverse event | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 2 | 5
Not completed — Other | 0 | 0 | 0 | 1
Not completed — Site Closed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg | Total
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (14.5) | 37.5 (10.4) | 46.3 (12.9) | 37.0 (11.5) | 39.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 7 | 10 | 35
  Male | 13 | 11 | 14 | 11 | 49

OUTCOME MEASURES:

1. Primary Outcome: Fold Change From Baseline in Fecal Calprotectin at Week 14
Description: The fold change from baseline in fecal calprotectin at Week 14, is the ratio of the measurement of fecal calprotectin at Week 14 to baseline measurement; this was calculated as the change from baseline in natural log transformed fecal calprotectin at Week 14.
Time Frame: Baseline, Week 14
Population: Modified Intent to Treat (mITT: all randomized participants who received greater than or equal to [>=] 1 dose study drug); Data as Observed (DAO: all mITT participants with all data needed for calculation of specified endpoint). "Number of Participants Analyzed" signifies participants in the mITT DAO population for specified endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: fold change
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 7 | 14 | 15 | 13
fold change | 0.41 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.29 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.79 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 1.24 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis.
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; Least squares (LS) mean = 0.41, 80% CI 2-sided [0.225 to 0.766] — LS mean and confidence interval (CI) were based on back log-transformation of those from the analysis of covariance (ANCOVA) model
Statistical Analysis 2: Comparison: Anrukinzumab 200 mg; Test type: Superiority or Other; LS mean = 0.29, 80% CI 2-sided [0.187 to 0.446] — LS mean and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 3: Comparison: Anrukinzumab 400 mg; Test type: Superiority or Other; LS mean = 0.79, 80% CI 2-sided [0.517 to 1.203] — LS mean and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 4: Comparison: Anrukinzumab 600 mg; Test type: Superiority or Other; LS mean = 1.24, 80% CI 2-sided [0.794 to 1.949] — LS mean and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 5: Comparison: Placebo vs Anrukinzumab 200 mg; P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.5320, ANCOVA; LS mean ratio = 0.70, 80% CI 2-sided [0.329 to 1.472] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 6: Comparison: Placebo vs Anrukinzumab 400 mg; P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.2700, ANCOVA; LS mean ratio = 1.90, 80% CI 2-sided [0.900 to 4.013] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 7: Comparison: Placebo vs Anrukinzumab 600 mg; P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.0666, ANCOVA; LS mean ratio = 3.00, 80% CI 2-sided [1.403 to 6.409] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Anrukinzumab
Description: Maximum concentration observed during the dosing interval (2 weeks for day 1, 4 weeks for week 12).
Time Frame: Pre-dose to end of the dosing interval after Day 1, Week 12
Population: All participants with evaluable pharmacokinetic (PK) results were included in PK population. PK samples with time deviation greater than (>) 20 percent (%) from nominal time were excluded from statistical summary and PK analysis. "Number of participants analyzed" = participants in PK population; "n" = evaluable participants at specified time point.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 20 | 20 | 21
nanogram/milliliter (ng/mL)
  Day 1 (n=19, 20, 20) | 54480 (15027) | 101200 (36239) | 182200 (64817)
  Week 12 (n=15, 16, 13) | 68270 (34360) | 121400 (43461) | 197600 (80647)

3. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Anrukinzumab
Description: Lowest concentration observed during the dosing interval (2 weeks for day 1, 4 weeks for week 12).
Time Frame: Pre-dose to end of the dosing interval after Day 1, Week 12
Population: All participants with evaluable PK results were included in PK population. PK samples with time deviation >20% from nominal time were excluded from statistical summary and PK analysis. "Number of participants analyzed" signifies participants in PK population; "n" signifies evaluable participants at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 20 | 20 | 21
ng/mL
  Day 1 (n=19, 20, 20) | 0.0000 (0.00000) | 42.45 (165.38) | 51.19 (201.57)
  Week 12 (n=15, 16, 13) | 13310 (8314.0) | 22350 (14281) | 31120 (16821)

4. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for Anrukinzumab
Description: Area under the plasma concentration curve from time zero to end of dosing interval (2 weeks) was reported.
Time Frame: Pre-dose, within 1 hour post-end of infusion on Day 1; Day 2, 4, 7, pre-dose on Week 2
Population: All participants with evaluable PK results were included in PK population. PK samples with time deviation >20% from nominal time were excluded from statistical summary and PK analysis. "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 19 | 20 | 20
nanogram*hour/milliliter (ng*hr/mL) | 8346000 (3622500) | 14670000 (6055800) | 24430000 (7657300)

5. Secondary Outcome: Plasma Decay Half-Life (t1/2) for Anrukinzumab
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: Within 1 hour post-end of infusion on Week 12; Week 14, 16, 18, 20, 22, 24, 26, 28, 30, 32
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 14 | 16 | 7
hours | 392.4 (99.107) | 470.5 (361.46) | 362.4 (111.18)

6. Secondary Outcome: Systemic Clearance (CL) for Anrukinzumab
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: Pre-dose, within 1 hour post-end of infusion on Week 12; Week 14, 16, 18, 20, 22, 24, 26, 28, 30, 32
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters/day
Arm/Group | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 15 | 16 | 13
liters/day | 0.2844 (0.15918) | 0.3090 (0.14268) | 0.3789 (0.23249)

7. Secondary Outcome: Volume of Distribution (Vz) for Anrukinzumab
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: Pre-dose, within 1 hour post-end of infusion on Week 12; Week 14, 16, 18, 20, 22, 24, 26, 28, 30, 32
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 14 | 16 | 7
liters | 5.726 (2.5057) | 9.704 (13.186) | 6.143 (2.1013)

8. Secondary Outcome: Fold Change From Baseline in Fecal Calprotectin at Week 2, 4, 8 and 12
Description: The fold change from baseline in fecal calprotectin at post-baseline visit, is the ratio of the measurement of fecal calprotectin at post-baseline visit to baseline measurement; this was calculated as the change from baseline in natural log transformed fecal calprotectin at post-baseline visit.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: mITT: all randomized participants who received >=1 dose study drug; DAO: all mITT participants with all data needed for calculation of specified endpoint. "Number of Participants Analyzed" signifies participants in mITT population; "n" signifies participants in mITT DAO population for specified time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: fold change
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21
fold change
  Fold Change at Week 2 (n=15, 17, 18, 13) | 0.70 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.81 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.71 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.77 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis.
  Fold change at Week 4 (n=14, 18, 19, 16) | 0.92 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.47 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.92 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.55 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis.
  Fold change at Week 8 (n=10, 16, 17, 16) | 0.78 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.36 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 1.14 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.52 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis.
  Fold change at Week 12 (n=9, 13, 14, 11) | 0.64 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.19 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.96 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.67 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis.
Statistical Analysis 1: Comparison: Placebo; Week 2: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.70, 80% CI 2-sided [0.466 to 1.048]
Statistical Analysis 2: Comparison: Anrukinzumab 200 mg; Week 2: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.81, 80% CI 2-sided [0.552 to 1.185]
Statistical Analysis 3: Comparison: Anrukinzumab 400 mg; Week 2: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.71, 80% CI 2-sided [0.488 to 1.027]
Statistical Analysis 4: Comparison: Anrukinzumab 600 mg; Week 2: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.77, 80% CI 2-sided [0.500 to 1.195]
Statistical Analysis 5: Comparison: Placebo; Week 4: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.92, 80% CI 2-sided [0.631 to 1.328]
Statistical Analysis 6: Comparison: Anrukinzumab 200 mg; Week 4: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.47, 80% CI 2-sided [0.339 to 0.655]
Statistical Analysis 7: Comparison: Anrukinzumab 400 mg; Week 4: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.92, 80% CI 2-sided [0.669 to 1.269]
Statistical Analysis 8: Comparison: Anrukinzumab 600 mg; Week 4: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.55, 80% CI 2-sided [0.388 to 0.779]
Statistical Analysis 9: Comparison: Placebo; Week 8: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.78, 80% CI 2-sided [0.454 to 1.331]
Statistical Analysis 10: Comparison: Anrukinzumab 200 mg; Week 8: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.36, 80% CI 2-sided [0.236 to 0.553]
Statistical Analysis 11: Comparison: Anrukinzumab 400 mg; Week 8: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 1.14, 80% CI 2-sided [0.757 to 1.722]
Statistical Analysis 12: Comparison: Anrukinzumab 600 mg; Week 8: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.52, 80% CI 2-sided [0.338 to 0.788]
Statistical Analysis 13: Comparison: Placebo; Week 12: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.64, 80% CI 2-sided [0.374 to 1.084]
Statistical Analysis 14: Comparison: Anrukinzumab 200 mg; Week 12: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.19, 80% CI 2-sided [0.122 to 0.297]
Statistical Analysis 15: Comparison: Anrukinzumab 400 mg; Week 12: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.96, 80% CI 2-sided [0.623 to 1.465]
Statistical Analysis 16: Comparison: Anrukinzumab 600 mg; Week 12: LS mean and CI were based on back log-transformation of those from the ANCOVA model; Test type: Superiority or Other; LS mean = 0.67, 80% CI 2-sided [0.411 to 1.076]
Statistical Analysis 17: Comparison: Placebo vs Anrukinzumab 200 mg; Week 2: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.7352, ANCOVA; LS mean ratio = 1.16, 80% CI 2-sided [0.663 to 2.021] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 18: Comparison: Placebo vs Anrukinzumab 400 mg; Week 2: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.9754, ANCOVA; LS mean ratio = 1.01, 80% CI 2-sided [0.586 to 1.753] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 19: Comparison: Placebo vs Anrukinzumab 600 mg; Week 2: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.8277, ANCOVA; LS mean ratio = 1.11, 80% CI 2-sided [0.609 to 2.008] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 20: Comparison: Placebo vs Anrukinzumab 200 mg; Week 4: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.0885, ANCOVA; LS mean ratio = 0.51, 80% CI 2-sided [0.313 to 0.846] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 21: Comparison: Placebo vs Anrukinzumab 400 mg; Week 4: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.9856, ANCOVA; LS mean ratio = 1.01, 80% CI 2-sided [0.617 to 1.644] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 22: Comparison: Placebo vs Anrukinzumab 600 mg; Week 4: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.1996, ANCOVA; LS mean ratio = 0.60, 80% CI 2-sided [0.361 to 1.000] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 23: Comparison: Placebo vs Anrukinzumab 200 mg; Week 8: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.1553, ANCOVA; LS mean ratio = 0.46, 80% CI 2-sided [0.233 to 0.926] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 24: Comparison: Placebo vs Anrukinzumab 400 mg; Week 8: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.4633, ANCOVA; LS mean ratio = 1.47, 80% CI 2-sided [0.748 to 2.882] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 25: Comparison: Placebo vs Anrukinzumab 600 mg; Week 8: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.4409, ANCOVA; LS mean ratio = 0.66, 80% CI 2-sided [0.335 to 1.316] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 26: Comparison: Placebo vs Anrukinzumab 200 mg; Week 12: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.0283, ANCOVA; LS mean ratio = 0.30, 80% CI 2-sided [0.150 to 0.598] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 27: Comparison: Placebo vs Anrukinzumab 400 mg; Week 12: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.4434, ANCOVA; LS mean ratio = 1.50, 80% CI 2-sided [0.758 to 2.970] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model
Statistical Analysis 28: Comparison: Placebo vs Anrukinzumab 600 mg; Week 12: P-value was calculated from ANCOVA model with terms for treatment group, baseline (in log scale); Test type: Superiority or Other; p = 0.9372, ANCOVA; LS mean ratio = 1.04, 80% CI 2-sided [0.510 to 2.141] — LS mean ratio and CI were based on back log-transformation of those from the ANCOVA model

9. Secondary Outcome: Total Interleukin-13 (IL-13) Level
Time Frame: Baseline, Day 2, 4, 7, Week 2, 4, 8, 12, 14, 16, 20, 24, 28, 32
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: picogram/milliliter
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21
picogram/milliliter
  Baseline (n=15, 21, 20, 19) | 0.6247 (0.97041) | 1.6231 (2.95190) | 1.2900 (2.07219) | 0.7525 (1.59494)
  Day 2 (n=21, 19, 17, 18) | 0.5980 (0.81335) | 3.6373 (4.69500) | 6.6673 (7.29515) | 5.0474 (4.97368)
  Day 4 (n=16, 16, 20, 15) | 0.7056 (1.29166) | 7.7698 (9.02951) | 12.3410 (11.84611) | 10.1349 (10.24068)
  Day 7 (n=7, 12, 9, 13) | 0.8991 (1.15883) | 15.6742 (34.90836) | 16.6700 (16.73533) | 11.3600 (16.79136)
  Week 2 (n=20, 21, 19, 19) | 0.7177 (0.98373) | 16.6373 (54.71391) | 17.7895 (18.53571) | 21.5021 (27.03784)
  Week 4 (n=18, 21, 19, 17) | 0.8949 (1.47538) | 15.1244 (43.76893) | 17.1853 (15.00105) | 8.7807 (5.39145)
  Week 8 (n=16, 18, 18, 15) | 0.7310 (1.09524) | 21.4964 (72.31269) | 16.8200 (15.47020) | 6.8027 (3.44810)
  Week 12 (n=12, 14, 17, 11) | 0.8925 (1.38386) | 19.3543 (52.00880) | 22.4335 (27.04635) | 6.8461 (4.19321)
  Week 14 (n=12, 14, 16, 13) | 1.0545 (1.15526) | 33.6697 (110.9546) | 20.0044 (37.36283) | 8.9492 (6.33317)
  Week 16 (n=10, 12, 12, 7) | 0.5054 (0.29982) | 15.0002 (40.41488) | 16.4423 (24.54910) | 3.7570 (2.91709)
  Week 20 (n=8, 15, 15, 8) | 1.5140 (1.82370) | 9.8396 (25.99516) | 7.4261 (8.00205) | 4.1745 (2.84220)
  Week 24 (n=10, 12, 12, 8) | 1.3300 (1.41349) | 3.0140 (3.23912) | 6.3665 (7.85116) | 3.0913 (1.99098)
  Week 28 (n=10, 12, 13, 8) | 1.2151 (2.23797) | 0.9936 (0.75719) | 2.8005 (2.67967) | 3.1724 (2.15647)
  Week 32 (n=9, 12, 13, 8) | 0.4727 (0.37875) | 1.0548 (0.80675) | 1.9379 (1.99196) | 2.4725 (2.54141)

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Week 32 that were absent before treatment or that worsened relative to pretreatment state. All causality AEs included SAEs as well as non-serious AEs, without regard to relationship to the study drug, which occurred during the trial.
Time Frame: Baseline up to Week 32
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21
participants
  AEs | 15 | 19 | 17 | 17
  SAEs | 4 | 4 | 2 | 4

11. Secondary Outcome: Number of Participants Who Discontinued From the Study Due to Adverse Events
Time Frame: Baseline up to Week 32
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21
participants | 4 | 5 | 1 | 5

12. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) and Neutralizing Antibody
Description: Neutralizing antibody was not analyzed as no participant had positive ADA samples.
Time Frame: Day 1, Week 4, 8, 12, 14, 16, 20, 24, 28, 32
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 21 | 21 | 21 | 21
participants
  Day 1 (n=18, 20, 19, 21) | 0 | 0 | 0 | 0
  Week 4 (n=17, 18, 20, 18) | 0 | 0 | 0 | 0
  Week 8 (n=15, 17, 18, 13) | 0 | 0 | 0 | 0
  Week 12 (n=14, 15, 17, 13) | 0 | 0 | 0 | 0
  Week 14 (n=13, 14, 15, 13) | 0 | 0 | 0 | 0
  Week 16 (n=10, 15, 14, 7) | 0 | 0 | 0 | 0
  Week 20 (n=11, 14, 15, 7) | 0 | 0 | 0 | 0
  Week 24 (n=10, 12, 14, 7) | 0 | 0 | 0 | 0
  Week 28 (n=8, 12, 13, 7) | 0 | 0 | 0 | 0
  Week 32 (n=10, 13, 15, 6) | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Clinical Response Rate at Week 14
Description: Clinical response rate is defined as percentage of participants with at least 3 point decrease from baseline in total Mayo score with at least 30% change along with 1 point decrease from baseline or absolute score of 0 or 1 in rectal bleeding. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, findings on flexible sigmoidoscopy [endoscopy] and physician's global assessment), each subscore is graded from 0 to 3 with the higher score indicating more severe disease activity.
Time Frame: Week 14
Population: mITT: all randomized participants who received >=1 dose study drug; DAO: all mITT participants with all data needed for calculation of specified endpoint. "Number of Participants Analyzed" signifies participants in the mITT DAO population for specified endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 12 | 15 | 16 | 13
percentage of participants | 41.67 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 60.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 50.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 15.38 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis.
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; percentage of participants = 41.67, 80% CI 2-sided [25.53 to 59.81] — CI was assessed by Wilson score method
Statistical Analysis 2: Comparison: Anrukinzumab 200 mg; Test type: Superiority or Other; percentage of participants = 60.00, 80% CI 2-sided [43.59 to 74.43] — CI was assessed by Wilson score method
Statistical Analysis 3: Comparison: Anrukinzumab 400 mg; Test type: Superiority or Other; percentage of participants = 50.00, 80% CI 2-sided [34.74 to 65.26] — CI was assessed by Wilson score method
Statistical Analysis 4: Comparison: Anrukinzumab 600 mg; Test type: Superiority or Other; percentage of participants = 15.38, 80% CI 2-sided [6.58 to 31.96] — CI was assessed by Wilson score method
Statistical Analysis 5: Comparison: Placebo vs Anrukinzumab 200 mg; Two-sided p-value was calculated by Fisher's exact test; Test type: Superiority or Other; p = 0.4495, Fisher Exact; percent difference = 18.33, 80% CI 2-sided [-6.13 to 39.98] — CI was assessed by Wilson score method
Statistical Analysis 6: Comparison: Placebo vs Anrukinzumab 400 mg; Two-sided p-value was calculated by Fisher's exact test; Test type: Superiority or Other; p = 0.7177, Fisher Exact; percent difference = 8.33, 80% CI 2-sided [-15.37 to 30.54] — CI was assessed by Wilson score method
Statistical Analysis 7: Comparison: Placebo vs Anrukinzumab 600 mg; Two-sided p-value was calculated by Fisher's exact test; Test type: Superiority or Other; p = 0.2016, Fisher Exact; percent difference = -26.28, 80% CI 2-sided [-46.45 to -3.15] — CI was assessed by Wilson score method

14. Other Pre Specified Outcome: Clinical Remission Rate at Week 14
Description: Clinical remission rate is defined as percentage of participants with a total Mayo score less than or equal to 2, with no individual subscore greater than 1 at post baseline visit. The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, findings on flexible sigmoidoscopy and physician's global assessment), each subscore is graded from 0 to 3 with the higher score indicating more severe disease activity.
Time Frame: Week 14
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 12 | 15 | 16 | 13
percentage of participants | 16.67 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 33.33 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 18.75 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | 0.00 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis.
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; percentage of participants = 16.67, 80% CI 2-sided [7.14 to 34.22] — CI was assessed by Wilson score method
Statistical Analysis 2: Comparison: Anrukinzumab 200 mg; Test type: Superiority or Other; percentage of participants = 33.33, 80% CI 2-sided [20.08 to 49.88] — CI was assessed by Wilson score method
Statistical Analysis 3: Comparison: Anrukinzumab 400 mg; Test type: Superiority or Other; percentage of participants = 18.75, 80% CI 2-sided [9.40 to 33.92] — CI was assessed by Wilson score method
Statistical Analysis 4: Comparison: Anrukinzumab 600 mg; Test type: Superiority or Other; percentage of participants = 0.00, 80% CI 2-sided [0.00 to 11.22] — CI was assessed by Wilson score method
Statistical Analysis 5: Comparison: Placebo vs Anrukinzumab 200 mg; Two-sided p-value was calculated by Fisher's exact test; Test type: Superiority or Other; p = 0.4082, Fisher Exact; percent difference = 16.67, 80% CI 2-sided [-5.33 to 35.76] — CI was assessed by Wilson score method
Statistical Analysis 6: Comparison: Placebo vs Anrukinzumab 400 mg; Two-sided p-value was calculated by Fisher's exact test; Test type: Superiority or Other; p = 1.0000, Fisher Exact; percent difference = 2.08, 80% CI 2-sided [-17.80 to 19.99] — CI was assessed by Wilson score method
Statistical Analysis 7: Comparison: Placebo vs Anrukinzumab 600 mg; Two-sided p-value was calculated by Fisher's exact test; Test type: Superiority or Other; p = 0.2200, Fisher Exact; percent difference = -16.67, 80% CI 2-sided [-34.22 to -1.95] — CI was assessed by Wilson score method

15. Other Pre Specified Outcome: Change From Baseline in Total Mayo Score at Week 14
Description: The Mayo score is a tool designed to measure disease activity for ulcerative colitis. The Mayo score ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, findings on flexible sigmoidoscopy [endoscopy] and physician's global assessment), each subscore is graded from 0 to 3 with the higher score indicating more severe disease activity.
Time Frame: Baseline, Week 14
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: unit on a scale
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 12 | 15 | 16 | 13
unit on a scale | -1.32 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | -2.28 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | -2.30 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis. | -0.79 [NA to NA] — Data is reported in the statistical analysis section because only 80% CI was calculated for this outcome measure as per planned analysis.
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority or Other; LS mean = -1.32, 80% CI 2-sided [-2.332 to -0.300]
Statistical Analysis 2: Comparison: Anrukinzumab 200 mg; Test type: Superiority or Other; LS mean = -2.28, 80% CI 2-sided [-3.190 to -1.374]
Statistical Analysis 3: Comparison: Anrukinzumab 400 mg; Test type: Superiority or Other; LS mean = -2.30, 80% CI 2-sided [-3.178 to -1.419]
Statistical Analysis 4: Comparison: Anrukinzumab 600 mg; Test type: Superiority or Other; LS mean = -0.79, 80% CI 2-sided [-1.761 to 0.190]
Statistical Analysis 5: Comparison: Placebo vs Anrukinzumab 200 mg; P-value was analyzed from ANCOVA model with terms for treatment group and baseline; Test type: Superiority or Other; p = 0.3639, ANCOVA; LS mean difference = -0.97, 80% CI 2-sided [-2.335 to 0.403]
Statistical Analysis 6: Comparison: Placebo vs Anrukinzumab 400 mg; P-value was analyzed from ANCOVA model with terms for treatment group and baseline; Test type: Superiority or Other; p = 0.3446, ANCOVA; LS mean difference = -0.98, 80% CI 2-sided [-2.320 to 0.355]
Statistical Analysis 7: Comparison: Placebo vs Anrukinzumab 600 mg; P-value was analyzed from ANCOVA model with terms for treatment group and baseline; Test type: Superiority or Other; p = 0.6285, ANCOVA; LS mean difference = 0.53, 80% CI 2-sided [-0.884 to 1.945]

16. Other Pre Specified Outcome: Number of Participants With Change From Baseline in Stool Frequency at Week 14
Description: Stool frequency is a sub score of Mayo score used to measure the disease activity of ulcerative colitis. The score for stool frequency ranges from 0 to 3, where higher score indicates more severe disease activity. Participant's score for stool frequency at Week 14 was specified as improved (decrease), no change and worsened (increase) compared to their baseline score.
Time Frame: Baseline, Week 14
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 12 | 15 | 16 | 13
participants
  Improvement | 4 | 7 | 7 | 3
  No Change | 8 | 4 | 8 | 6
  Worsening | 0 | 4 | 1 | 4

17. Other Pre Specified Outcome: Number of Participants With Change From Baseline in Rectal Bleeding at Week 14
Description: Mayo score is used to measure the disease activity of ulcerative colitis. Rectal bleeding is a sub score of Mayo score. The score for rectal bleeding ranges from 0 to 3, where higher score indicates more severe disease activity. Participant's score for rectal bleeding at Week 14 was specified as improved (decrease), no change and worsened (increase) compared to their baseline score.
Time Frame: Baseline, Week 14
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 12 | 15 | 16 | 13
participants
  Improvement | 4 | 8 | 7 | 5
  No Change | 6 | 6 | 6 | 7
  Worsening | 2 | 1 | 3 | 1

18. Secondary Outcome: Number of Participants With Change From Baseline in Endoscopic Subscore at Week 14
Description: Mayo score is used to measure the disease activity of ulcerative colitis. Endoscopy or flexible sigmoidoscopy is a sub score of Mayo score. The score for endoscopic subscore ranges from 0 to 3, where higher score indicates more severe disease activity. Participant's score for endoscopy or flexible sigmoidoscopy at Week 14 was specified as improved (decrease), no change and worsened (increase) compared to their baseline score.
Time Frame: Baseline, Week 14
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Number analyzed (Participants) | 12 | 15 | 16 | 13
participants
  Improvement | 6 | 8 | 11 | 2
  No Change | 3 | 5 | 5 | 11
  Worsening | 3 | 2 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Anrukinzumab 200 mg | Anrukinzumab 400 mg | Anrukinzumab 600 mg
Serious Adverse Events (participants affected / at risk) | 4/21 | 4/21 | 2/21 | 4/21
Other Adverse Events (participants affected / at risk) | 12/21 | 18/21 | 13/21 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Anrukinzumab 200 mg (N=21) | Anrukinzumab 400 mg (N=21) | Anrukinzumab 600 mg (N=21)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 3 | 2 | 1 | 3
Cholangitis sclerosing (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=21) | Anrukinzumab 200 mg (N=21) | Anrukinzumab 400 mg (N=21) | Anrukinzumab 600 mg (N=21)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 4 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Vision blurred (Eye disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 2 | 3
Colitis ulcerative (Gastrointestinal disorders) | 3 | 7 | 5 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Chest pain (General disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 2 | 1
Oedema peripheral (General disorders) | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 1 | 0
Influenza (Infections and infestations) | 2 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 3 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 4 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.